CLINICAL TRIAL: NCT05845749
Title: A Proof of Concept Study to Evaluate the Safety and Efficacy of Voxzogo (Vosoritide) for the Treatment of Growth Deficits in MPS IVA and VI
Brief Title: Safety and Efficacy of Voxzogo for Growth Deficits in MPS IVA and VI
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Paul Harmatz, MD, Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-37966
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: MPS IVA; MPS VI
Keywords: Growth; Vosoritide; Children; Height; Voxzogo
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidosis VI | interventions — vosoritide

STUDY DESIGN:
Intervention Model Description: This is a 24 week natural history study followed by a 48 week open label single arm intervention with vosoritide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosoritide (Other): This is a single arm open label study of daily SQ dose of vosoritide
  Interventions: Drug: Vosoritide Injection [Voxzogo]

INTERVENTIONS:
Drug: Vosoritide Injection [Voxzogo] — Vosoritide will be given via a once daily subcutaneous injection at a dose of 15 ug/kg/day, at approximately the same time each day when feasible. Vosoritide will be supplied to the subject as 0.4 mg vial, 0.56 mg vial or 1.2 mg vials to be reconstituted with sterile water up to 0.8 mg/mL or 2 mg/mL concentrations for injection. The volume to be administered (injection volume) will be based on the subject's body weight and the concentration of vosoritide. All supplies will be provided to the subject for home based administration after training at the study site.
  Other Names: Vosoritide; BMN111

SUMMARY:
This is a Phase I/II, single arm, open label study of vosoritide therapy provided subcutaneously at 15 ug/kg/day for 48 weeks to 6 patients with MPS IVA or VI. Prior to enrollment in the interventional arm of study, subjects will be followed for a minimum of 24 weeks to gather information on safety profiles and determine annualized growth velocity. The primary study endpoint is the determination of safety and tolerability of daily vosoritide treatment in MPS. Exploratory endpoints include changes in linear and segmental growth as well as biomarkers of growth and bone metabolism.

DETAILED DESCRIPTION:
The investigators propose to conduct a single arm phase I/II study of Vosoritide (also called VOXZOGO® and BMN111) in 6 pediatric patients with mucopolysaccaridosis (MPS) types IVA and VI; 3 patients with each disease. This will be a single center study performed at UCSF Children's Hospital, Oakland, under the direction of Dr. Paul Harmatz, Professor in Residence in the Department of Pediatric Gastroenterology.

Mucopolysaccharidoses (MPS) are a group of ultra rare genetic lysosomal storage diseases caused by deficiency in various enzymes responsible for the breakdown of glycosaminoglycans (GAGs), leading to progressive accumulations of GAGs in the tissues and organs. Patients with MPS have severe growth deficits and growth-related decreased quality of life. In this study, the MPS disorders which have the most severe growth deficits will be the focus, MPS IVA and VI.

Enzyme replacement therapies (ERT) have been developed and approved for use in MPS. Though ERT has improved functional outcomes it does not lead to complete reversal of disease progression. Patients maintained on ERT continue to experience significant growth deficits.

Vosoritide, a CNP analog and recently approved FDA drug, has been shown to improve linear growth in patients with achondroplasia.

This proposal is for a Phase I/II, single arm, open label study of vosoritide therapy provided subcutaneously at 15 ug/kg/day for 48 weeks to 6 patients with MPS IVA or VI. Subjects will be included if they are > 5 years and < 10 years, Tanner pubertal stage 1 with a height Z-score of <-2.0 or less than 2 cm change in height velocity over the year prior to screening. Prior to enrollment in the interventional arm of study, subjects will be followed for a minimum of 24 weeks to gather information on safety profiles and determine pre-treatment (baseline) annualized growth velocity. The primary study endpoint is the determination of safety and tolerability of daily vosoritide treatment in MPS. Segmental growth, other functional assessments, inflammation, and bone/collagen markers, as well as quality of life will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 5 years and < 10 years
* Tanner stage 1
* Clinical Diagnosis of MPS IVA or VI

Subjects will be stratified into 2 groups:

* MPS IVA (3 patients)
* MPS VI (3 patients)

  * MPS Diagnosis Confirmed by either:

    1. Demonstration of 2 pathogenic or likely pathogen mutations (or homozygous for single mutation) and elevated GAG (either before or during ERT treatment), OR
    2. Demonstration of diagnostic enzyme deficiency, elevated GAG (either before or during ERT treatment), and a normal second sulfatase
  * Currently receiving ERT [elosulfase alfa (Vimizim®) or galsulfase (NAGLAZYME®)] for minimum of 12 months prior to study entry
  * HSCT greater than 3 years before entry
  * Height Z-score <-2.0 or less than 2 cm change in height velocity over the last 1 year
  * Willing to consent to the study and comply with all study procedures and assessments
  * Able to stand independently without hand support for minimum of one minute
  * Guardians able to successfully administer investigational drug daily/SQ

Exclusion Criteria:

* ERT naïve
* Poor compliance with ERT (<75% in 6 month period)
* Diagnosis with growth hormone deficiency (defined by IGF-1 SDS <-1.0 according to age, gender and tanner stage)
* Hypothyroidism, untreated (TSH >4.0 mU/L)
* Receiving or has received growth hormone therapy, IGF-1 therapy, anti-TNF alpha therapy, angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, diuretics, beta-blockers, calcium channel blockers, cardiac glycosides, systemic anticholinergic agents, any medication that may impair or enhance compensatory tachycardia, diuretics or other drugs known to alter renal or tubular function within the previous 6 months.
* Receiving or has previously received a GnRH analog (e.g. leuprolide acetate, histrelin)
* History of malignancy
* History of chronic inflammatory condition not related to MPS
* History of conditions/medical therapies that might affect the interpretation of growth results such as anemia, celiac disease, diabetes, inflammatory bowel disease, and cystic fibrosis
* QTC (Fridericia) > 450 msec
* Malnutrition (BMI <5th percentile)
* History of gene therapy
* Concurrent participation on an investigational drug trial
* Investigational drug washout minimum of 5 half-lives of the drug or 1 month whichever is longer
* Previous or current treatment with the investigational drug (vosoritide)
* Known or suspected allergy to the investigational drug (vosoritide)
* Bone fracture within the previous 6 months
* Skeletal surgery within the previous 6 months, or anticipated significant surgery (in the view of the investigator) during course of the study
* Any history of bone lengthening surgeries or spine fixation surgery
* Spine curvature (scoliosis) on previous x-ray greater than 25 degrees
* Untreated severe sleep apnea
* History of chronic renal insufficiency, defined previously as an eGFR <60 mL/min/1.73m2
* Illness that could affect blood pressure / orthostatic problems
* Treated with medications known to affect QC/QTc
* LV Ejection fraction <40%; LVEF=[SV/EDV] x100 (American Society Echocardiography)
* Treated with chronic oral steroids in previous 6 months
* Mean SpO2 of < 92% at baseline, taken from average of 3 measurements in each hand
* Concurrent disease or condition that in the view of the investigator, would interfere with study participation or safety evaluations, for any reason.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of adverse events while treated with vosoritide | 48 weeks
  Incidence of treatment-emergent adverse events as assessed by the evaluation of vital signs, pulse oximetry, pulmonary function, ECG (cardiac arrhythmia), ECHO (doppler of aortic velocity for stenosis, aortic valve area, and qualitative assessment of aortic valve thickness), spinal X-rays (worsening scoliosis, lordosis or kyphosis), standing lower extremity X-rays (worsening of genu valgum), decrease in six-minute walk distance and linear and segmental growth for determination of excessive or disproportionate growth. All safety assessments will be performed at a minimum at the beginning of the intervention (Visit 1) and the end of the intervention (Visit 3) in patients with MPS IVA and VI

SECONDARY OUTCOMES:
Change in height velocity while treated with vosoritide | 72 weeks
  Explore the change from baseline (0-24 weeks pre-intervention) in age-sex annualized height velocity after 48 weeks of daily subcutaneous vosoritide therapy in patients with MPS IVA and VI

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harmatz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No